CLINICAL TRIAL: NCT01490164
Title: An Observational Prospective Study of Transfusion Requirements During Spinal Surgery for Severe Scoliosis
Brief Title: Transfusion Requirements During Spinal Surgery for Severe Scoliosis
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anesthesia, Department of Anesthesia/Investigator initiated, Rutgers, The State University of New Jersey
Other Study IDs: 0120090203
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- scoliosis: young adults requiring surgical correction

SUMMARY:
Corrective surgery for scoliosis can result in prolonged operating room time and significant blood loss. The investigators goal is to determine what the transfusion requirements are for young adults undergoing spinal surgery for scoliosis and what other intra-operative factors influence the amount of blood and blood products used. The investigators will used the information obtained to improve the management of patients undergoing corrective surgery for scoliosis.

DETAILED DESCRIPTION:
Data collected prior to surgery will include patients' past medical history, hemoglobin concentration, INR, MCV, gender, age and weight.

Immediately prior to surgery, but after induction of anesthesia, subjects will have another complete blood count drawn to assess preoperative hemoglobin/hematocrit concentrations. This is customarily done to establish a baseline. During surgery patient's core temperature, hemoglobin, hematocrit levels, estimated blood loss, Central Venous Pressure, blood pressure, heart rate, cell saver, the amount of irrigation fluid, colloid, crystalloid, blood and blood products will be recorded hourly throughout surgery. All of the data collection described is standard in these types of cases.

Patients will be transfused allogenic blood if hemoglobin levels fall below 8.0 g/dL or patients present with clinical signs/symptoms of hypovolemia (hypotension, tachycardia). Data collection concerning allogenic blood transfusion will include intraoperative transfusion rate, volume of transfused units per patient and transfusion index. Surgical intervention data regarding the extent of the surgical procedure will be collected: the number of curves, the curve magnitude, type of instrumentation required, the number of levels fused and the fluoroscopy time. The placement and type of wound drains and their .respective outputs will be noted. Preoperative and postoperative curve magnitude will be documented as well as instrumentation used to facilitate curve correction. The number of levels fused will be documented.

Hemoglobin and hematocrit levels will be noted at several intervals post operatively (24 hours, 48 hours and last result prior to discharge) and further transfusion requirement will be recorded. The length of Intensive Care Unit stay and the length of hospital stay will be noted. Regarding surgical procedure all patients will be operated on by the same surgical team, under standardized anesthesia, total intravenous anesthesia (TIVA), and postoperative analgesia. Data will be expressed as percentages or as a mean +/- SD. T-test analysis will be used for comparison for quantitative variables and a p value < 0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing surgical correction of scoliosis

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all patients undergoing surgical correction of scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
transfusion requirements | 0-72 hours
  number of blood transfusion subject required from surgical start time to 72 hours post op

SECONDARY OUTCOMES:
vertebral levels fused | intraoperatively
  number of vertebral levels fused

OTHER OUTCOMES:
operative time | time in OR
  surgical start and finish times
ICU stay | days
  number of stays subject stays in ICU
hospital days | days
  number of days until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Patel, MD, Principal Investigator — UMDNJ/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States